CLINICAL TRIAL: NCT00929786
Title: Measurement of Drug Levels and Their Correlation With Hepatotoxicity During Antituberculosis Treatment
Brief Title: Anti-tuberculosis (TB) Drug Levels and Hepatotoxicity
Status: Completed | Type: Observational
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Dr. S K Sharma, Department of Medicine, AIIMS, New Delhi-110029
Other Study IDs: SKS/DIH/01; sksharma@aiims.ac.in
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Hepatitis; Tuberculosis
Keywords: Plasma levels isoniazid rifampicin pyrazinamide
MeSH Terms: conditions — Hepatitis; Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 2: Cases - those patients who develop DIH while on regular treatment with anti-TB drugs.
  Controls - patients who do not develop DIH while on regular treatment with anti-TB drugs.

SUMMARY:
The purpose of this study is to evaluate plasma levels of hepatotoxic anti-tuberculous drugs (isoniazid, rifampicin, pyrazinamide plus significant metabolites) among patients on antituberculosis treatment (ATT) and compare the same among those who develop drug induced hepatitis on follow up versus those who do not.

DETAILED DESCRIPTION:
Tuberculosis (TB) is a major health problem in both the developing and developed countries because of its resurgence in the immunosuppressed patients. World Health Organization (WHO) in 1993 declared tuberculosis to be a 'global emergency' with more than a third of the world's population infected. Globally 8.9 million new cases of tuberculosis occur annually, of which 1.8 million (20%) occur in India.

Short-course chemotherapy containing isoniazid (INH), rifampicin (RMP) and pyrazinamide (PZA) has proved to be highly effective in the treatment of tuberculosis. One of its adverse effects is hepatotoxicity. It is the most common side effect leading to interruption of therapy. It is associated with mortality of 6-12% if these drugs are continued even after the onset of symptoms. Risk of hepatotoxicity is increased when these drugs are combined.

The time interval between the start of anti-TB drugs and appearance of hepatotoxicity varies from 3 to 135 days. In most cases hepatitis is evident within three months of start of antituberculosis treatment (ATT).

The pathogenesis of drug-induced hepatotoxicity (DIH) is still not entirely clear for most anti TB drugs including rifampicin. Hypersensitivity is a definite possibility Rifampicin induced hepatitis has been postulated to occur as a part of systemic allergic reaction and, due to unconjugated hyperbilirubinaemia as a result of competition with bilirubin for uptake at hepatocyte plasma membrane. DIH caused by rifampicin occurs earlier as compared to isoniazid. While a dose related toxicity may exist, a direct correlation between serum drug levels and hepatotoxicity has not been well reported. Thus the clinical relevance of therapeutic monitoring of serum rifampicin concentrations in managing DIH is still being explored.

Present study done to observe serum rifampicin, isoniazid, pyrazinamide level in patients on ATT and to compare it retrospectively between patients who develop drug induced hepatitis vs those who do not.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed to be suffering from CatI/CatIII tuberculosis by a physician
2. Age: 16-65 years
3. Patient having normal baseline Liver function (AST/ALT1 < 50/50, serum bilirubin < 1.5 mg/dl)

Exclusion Criteria:

1. Patients receiving any other drug known to be metabolized by liver by cytochrome P450 3A4 or P-glycoprotein
2. Patients diagnosed to have acute viral hepatitis A, B, C, or E or carrier for HBV & HCV
3. Known HIV positive patients
4. Presence of chronic liver disease or renal insufficiency
5. Concomitant administration of other potential hepatotoxic drugs (methotrexate, phenytoin, valproate)
6. Chronic alcoholics who consume > 48 g of alcohol/day for at least one year
7. Pregnant women
8. Subjects not willing to participate
9. Known patients with malabsorption or drug abuse

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects: Patients with diagnosis of CatI/CatIII Tuberculosis attending the out-patient department of the All India Institute of Medical Sciences, New Delhi, will form the study population.
  Cases - those patients who develop DIH while on regular treatment with anti-TB drugs Controls - age, sex matched patients who do not develop DIH while on regular treatment with anti-TB drugs
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2007-11; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of plasma levels of isoniazid, rifampicin, pyrazinamide among cases and controls | 20 months

SECONDARY OUTCOMES:
Evaluation of plasma levels of any significant metabolites among cases and controls | 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Surendra K Sharma, MD,Ph.D, Principal Investigator — All India Institute of Medical Sciences, New Delhi-110029, India
Locations (2):
- India (2):
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, New Delhi, New Delhi